CLINICAL TRIAL: NCT03637478
Title: Enhancing Systems of Care: Supporting Families and Improving Youth Outcomes
Acronym: E-SOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Responsible Party: Principal Investigator, Katherine Grimes MD, Director, Children's Health Initiative, Harvard Medical School (HMS and HSDM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CHR-IRB-1062/04/17
Record Dates: First submitted 2018-07-19; First posted 2018-08-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Pediatric Mental Health Services

STUDY DESIGN:
Intervention Model Description: The E-SOC Model consists of the delivery of intensively integrated clinical care within pediatrics, combined with community-based parent support from family support specialists. Innovations include child mental health specialists joining the pediatrics team for "huddles", psychiatry notes shared with pediatricians via the Electronic Medical Records and active inclusion of pediatricians in pre-evaluation discussions with the E-SOC Team and post-evaluation recommendations for the families. In addition, the E-SOC model includes active communication with school personnel, child welfare, and community-based resources, when needed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enhanced Systems of Care Team (Experimental): The four intervention sites have been selected based on their size: taken together, their pediatric populations comprise over 80% of the total number of children receiving care at Cambridge Health Alliance. At the four intervention sites, the study will involve: 1) an integrated child mental health assessment done by the E-SOC team within primary care, 2) active follow-up, collaboration with specialty providers and support to families, 3) School, child welfare and other community linkages as appropriate.
  Interventions: Behavioral: Enhanced Systems of Care Team

INTERVENTIONS:
Behavioral: Enhanced Systems of Care Team — E-SOC team will be increasing connections between clinical care and community partners, such as schools, juvenile justice and child-serving state agencies, to reduce disparities in access to mental health/substance use evaluation and treatment. All aspects of the care continuum will be provided in a culturally and linguistically competent manner, with child and family-driven care planning. Overall goals are: earlier identification of mental health needs including child trauma; increased treatment access and adherence; care delivered in least restrictive settings; care experience reflecting active youth and family engagement; program sustainability and replicability.

SUMMARY:
The aim of the study is to improve access to child mental health and substance abuse (MH/SA) care by expanding primary care screening and increasing availability of timely mental health evaluation and treatment.

DETAILED DESCRIPTION:
This is a quasi-experimental, longitudinal study. Identified youth and families will receive the intervention within the four study site clinic locations. Comparison group families will receive usual care. Each primary care study site will have designated Family Support Specialist, Clinical Care Manager and Child Psychiatry resources. The intervention includes an integrated care consultation which combines diagnostic evaluation, family assessment, and multi-disciplinary, team-based treatment recommendations, with follow-up community linkages and support, as indicated.

ELIGIBILITY:
Inclusion Criteria:

* Must be between ages 0 to 17.5 years
* Referred by primary care physician at one of these Cambridge Health Alliance clinics: Windsor Street Care Center, Broadway Care Center, Everett Care Center, Malden Family Medicine Center
* Referred youth must have a caregiver (a parent of guardian) who agrees to participate in the assessment and treatment process

Exclusion Criteria:

* 17.6 years or older

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Access to child mental health and substance abuse (MH/SA) care | Comparative analysis of access to care trends (0-6 months)
  Service Use Data from Electronic Health Records and Claims for intervention group versus controls
Engagement in child mental health and substance abuse (MH/SA) treatment | Comparative analysis of service use trends (6-12 months)
  Service Use Data from Electronic Health Records and Claims for intervention group versus controls

SECONDARY OUTCOMES:
Family Care Experience | Analysis of baseline and follow-up family perceptions of care (baseline collected at enrollment, follow-up assessments collected at 6 months and 12 months)
  Qualitative assessment of family perceptions of care using the Family Professional Partnership Scale (FPPS). The anchors of items rated on satisfaction are rated on a 5-point likert scale, where 1 = very dissatisfied, 3 = neither satisfied nor dissatisfied, and 5 = very satisfied wherein the higher the value represents a better outcome.
Changes in Children's Global Assessment Scale (CGAS) Score | Comparative analysis of baseline and follow-up clinical functioning scores (baseline collected at enrollment, follow-up assessments collected at 6 months and 12 months)
  Measurement of clinical functioning using Children's Global Assessment Scale (CGAS). Trends from baseline to 6 months and 12 months will be examined to identify improvement, decline, or no change in clinical functioning.The CGAS measure provides a single global rating only, on scale of 0-100, where scores below 60 indicate clinical need.
Changes in Child and Adolescent Functional Assessment Scale (CAFAS) Score | Comparative analysis of baseline and follow-up clinical functioning scores (baseline collected at enrollment, follow-up assessments collected at 6 months and 12 months)
  Measurement of clinical functioning using Child and Adolescent Functional Assessment Scale (CAFAS). Trends from baseline to 6 months and 12 months will be examined to identify improvement, decline, or no change in clinical functioning. The CAFAS measure indicates the level of clinical functioning, on a scale of 0-140, where scores above 40 indicate clinical need.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E Grimes, MD, MPH, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT03637478/ICF_000.pdf